CLINICAL TRIAL: NCT06801236
Title: A Phase 1 Study to Assess the Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of ACE-232 in Patients With Metastatic Castration-Resistant Prostate Cancer (CRPC)
Brief Title: Phase 1 Study of ACE-232 to Treat Patients With Metastatic Castration-Resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Acerand Therapeutics (Hong Kong) Limited (Industry)
Responsible Party: Sponsor
Organization: Acerand Therapeutics Limited (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-232-001
Record Dates: First submitted 2025-01-19; First posted 2025-01-30 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer (Adenocarcinoma); mCRPC (Metastatic Castration-resistant Prostate Cancer)
Keywords: ACE-232; castration-resistant prostate cancer; CRPC; Hormone Antagonists; Hormone Substitutes; Antineoplastic Agents; Prostatic Neoplasms; Castration-Resistant; prostate cancer; CYP11A1
MeSH Terms: conditions — Prostatic Neoplasms; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACE-232 (Experimental)
  Interventions: Drug: ACE-232 tablets

INTERVENTIONS:
Drug: ACE-232 tablets — ACE-232 tablets will be administered orally daily as a continuous regimen together with Dexamethasone and Fludrocortisone. Subjects will continue to receive study treatment until PD as judged by local investigator review, development of unacceptable toxicity, or withdrawal of consent.

SUMMARY:
This is an open label, phase I, multi-center study aiming to assess the safety and tolerability in patients with metastatic castration resistant prostate cancer (mCRPC).

DETAILED DESCRIPTION:
The study consists of two parts, Phase 1A dose escalation and Phase 1B dose optimization. Phase 1A aims to assess the safety, tolerability, pharmacokinetic (PK) profile, and changes in pharmacodynamic (PD) markers in patients treated with ACE-232, and to determine the maximum tolerated dose (MTD), if applicable. In Phase 1B, patients with AR gene alterations will be treated at two different dose levels to establish the recommended Phase 2 dose (RP2D).

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Metastatic Castration-resistant Prostate Cancer with ongoing androgen - deprivation therapy (ADT) or have bilateral orchiectomy
* Difficult to treat or intolerant to standard treatment (post at least 1 line of NHA and taxane-based chemo in mHSPC or mCRPC), suitable for investigational treatment;
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Has a life expectancy of at least 6 months
* Adequate organ function and bone marrow function

Exclusion Criteria:

* Receiving any anti-cancer drugs or other treatment, major surgery, extensive radiation therapy, or local radiation therapy within protocol-defined wash-out period;
* Concomitant use of medications or herbal supplements known to be moderate to strong CYP3A4 inhibitors/inducers, or P-gp inhibitors, known to prolong the QT interval.
* Any previous treatment-related toxicities have not recovered.
* Spinal cord compression or known brain metastases or leptomeningeal carcinomatosis.
* Severe cardiovascular disorders.
* Known gastrointestinal (GI) disorder or GI procedure
* History of gastric and duodenal perforation.
* History of pituitary dysfunction.
* Poorly controlled diabetes mellitus.
* Active or uncontrolled autoimmune disease
* Active infections, or a known history of HIV infection, or a known active hepatitis B or C, or a known active tuberculosis.
* Other malignancies requiring treatment within 3 years prior to the first dose of study drug
* Known allergy or hypersensitivity to any of the excipients of ACE-232.
* Has other medical conditions that at the discretion of the investigator interfere with safety or efficacy evaluation, or treatment compliance.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 67 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients experiencing adverse events (AEs)/serious adverse events (SAEs) | From time of information consent to 30 days post last dose, up to approximately 37 months
  Number of patients with incidence of adverse events and with serious adverse events including changes from baseline in laboratory parameters, vital signs, ECGs, and physical examination, etc.
Number of patients experiencing dose limiting toxicity (DLT), as defined in the protocol | From the first dose of ACE-232 on Cycle 1 Day 1 up to and including the planned end of Cycle 1 (at the end of 28 days)
  A DLT is defined as any toxicity events related to ACE-232 that occur from the first dose of study treatment until the planned end date of Cycle 1 (DLT assessment period), meeting the criteria specified in protocol.
Recommended Phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) | Up to approximately 37 months
  RP2D will be finally determined by the SMC and sponsor based on all data from the dose escalation module and backfill module, as well as the exposure-response relationship evaluated (if available). MTD is defined as the maximum dose level at which ≤1 patient have DLTs during the DLT observation period, and it should be determined with 6 evaluable patients.

SECONDARY OUTCOMES:
Pharmacokinetics characterization by using Area under the plasma concentration versus time curve (AUC) | Up to approximately 37 months
  To determine the pharmacokinetics (PK) using AUC of ACE-232 after a single dose and at steady state after multiple doses.
Pharmacokinetics characterization by using Maximum concentration (Cmax) | Up to approximately 37 months
  To determine the pharmacokinetics (PK) using Cmax of ACE-232 after a single dose and at steady state after multiple doses
Prostate Specific Antigen (PSA) response | Up to approximately 37 months
  PSA response is defined as PSA decline of 30% and 50% from baseline at any time point
Objective Response Rate (ORR) | Up to approximately 37 months
  ORR is defined as a complete response (CR) or partial response (PR), as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) and Prostate Cancer Working Group Criteria 3 (PCWG3 criteria), in patients with measurable disease at baseline.
Duration of Response (DoR) | Up to approximately 37 months
  DOR is defined, for patients with an objective response, as the time from first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or death due to any cause.
Radiographic Progression Free Survival (rPFS) | Up to approximately 37 months
  rPFS is defined as the time from the first dose of ACE-232 to the first documented disease progression by either RECIST progression and/or progression on bone scan by PCWG3 or death due to any cause, whichever occurs first.
Overall Survival (OS) | Up to approximately 37 months
  OS is defined as the time from the first dose of ACE-232 to the date of death due to any cause.
Blood concentration of steroid hormone | Up to approximately 37 months
  To determine the blood concentration of steroid hormones at various timepoints and change from baseline

OTHER OUTCOMES:
Gene aberrations | Up to approximately 37 months
  To determine the gene aberrations in circulating tumor DNA (ctDNA), and its association with tumor response or resistance to ACE-232

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California San Diego, Moores Cancer Center, La Jolla, California
  - Moffitt Cancer Center, Tampa, Tampa, Florida
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Harvard Medical School-Massachusetts General Hospital, Boston, Massachusetts
  - M Health Fairview Clinics and Surgery Center, Minneapolis, Minnesota
  - Xcancer (Urology Cancer Center), Omaha, Nebraska
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
No IPD sharing plan at this moment, which might be changed during the study process or when the results come out.